CLINICAL TRIAL: NCT05318339
Title: Open-label, Single-arm Phase II Study of Trastuzumab and Pyrotinib Combination Regimen in HER2 Positive Locally Advanced or Metastatic Urothelial Carcinoma Refractory to Standard Therapies
Brief Title: A Study of Trastuzumab and Pyrotinib in HER2 Positive Locally Advanced or Metastatic Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aiping Zhou, Vice director of Department of Medical Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC3398
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Carcinoma, Transitional Cell; HER-2 Gene Amplification
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Trastuzumab; pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab + Pyrotinib (Experimental): Patients receive a loading dose of trastuzumab IV over 90 minutes on day 1 of week 1. For all subsequent doses, patients receive trastuzumab IV over 30 minutes every three weeks.
  Meanwhile, patients also receive pyrotinib 400mg PO daily. Treatment may continue till unacceptable toxicity or disease progression occurs.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — A loading dose of trastuzumab 8mg/kg IV over 90 minutes will be administrated on day 1 of week 1.
  For all subsequent doses, trastuzumab 6mg/kg IV over 30 minutes will be administrated every three weeks.
  Pyrotinib 400mg PO daily will be administrated at the same time.
  Other Names: Pyrotinib

SUMMARY:
A open-label, single-arm, phase II trial to study was designed to evaluate the effectiveness and safety of trastuzumab and pyrotinib in treating HER2 positive patients who have previously treated, locally advanced, or metastatic urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form
* Locally advanced or metastatic histologically confirmed transitional cell carcinoma of the urothelium, including the bladder, urethra, ureter, or renal pelvis
* 18 years and older
* HER2 expression (3+ or 2+) as determined by immunohistochemistry or gene amplification by fluorescent in situ hybridization
* Relapsed from or failed at least one prior standard systemic chemotherapy regimen, including immunotherapy, HER2 ADC durgs, and chemothearpy containing cisplatin, carboplatin, paclitaxel, docetaxel, or gemcitabine
* At least 1 measurable lesion could be evaluated by RECIST v1.1
* Performance status: ECOG 0-1
* Life expectancy more than 12 weeks
* Ejection fraction at least 50% (or lower limit of normal) by echocardiogram
* Good organ function:

Blood routine: hemoglobin ≥80g/L, neutrophil ≥1.5×10^9/L, platelet ≥75×10^9/L; Renal function: creatinine≤1.5×upper limit of normal (UNL) or creatinine clearance ≥50ml/min; Liver function: total bilirubin (TBIL)≤1.5×upper limit of normal (UNL); ALT≤2.5×UNL, AST≤2.5×UNL, ALT≤5×UNL and AST≤5×UNL for patients with liver metastasis

Exclusion Criteria:

* Have received trastuzumab or pyrotinib treatment in the past
* Known to have allergic reactions to any ingredients or excipients of experimental drugs
* Radiotherapy, RFA, interventional therapy or surgery were performed within 28 days before the first medication (except for previous diagnostic biopsy)
* Other active malignant tumors, excluding those who have been disease free for more than 5 years or in situ cancer considered to have been cured by adequate treatment
* Clinically significant ascites
* Brain metastasis or meningeal metastasis with neurological symptoms
* Diabetes was not controlled, defined as HbA1c > 7.5% after anti-diabetic drugs or hypertension was not controlled, defined as systolic / diastolic blood pressure > 140 / 90 mmHg after antihypertensive drug
* Myocardial infarction, severe/unstable angina, New York Heart Association (NYHA) class III or IV congestive heart failure in the past 12 months
* Known to be infected with human immunodeficiency virus (HIV), have acquired immunodeficiency syndrome (AIDS) related diseases, have active hepatitis B or hepatitis C
* Pregnant or nursing
* May increase the risk associated with participation in the study or administration of the study drug or mental illness that may interfere with the interpretation of research results
* There are other serious diseases that the researchers believe patients cannot be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  Objective response rate as assessed by RECIST criteria

SECONDARY OUTCOMES:
OS | From date of initiation of treatment to date of death due to any cause, assessed up to 2 years
  Overall survival
PFS | From date of initiation of treatment to date of progression or death due to any cause, whichever occurs first, assessed up to 2 years
  Progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China